CLINICAL TRIAL: NCT05329623
Title: A Phase 1, Open-label, Single-dose, Multi-center, Parallel Group Study to Evaluate the Pharmacokinetics of JDQ443 in Participants With Mild, Moderate or Severe Hepatic Impairment Compared to Matched Healthy Control Participants.
Brief Title: A Phase 1 Study to Evaluate the Pharmacokinetics of JDQ443 in Participants With Hepatic Impairment Compared to Matched Healthy Control Participants.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CJDQ443B12103
Record Dates: First submitted 2022-03-29; First posted 2022-04-15 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Small Cell Lung Carcinoma
Keywords: JDQ443; pharmacokinetics; Child-Pugh classification; hepatic impairment
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — JDQ443

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Normal hepatic function (Experimental): Matched healthy participants with normal hepatic function
  Interventions: Drug: JDQ443
- Mild hepatic impairment (Experimental): Mild hepatic impaired participants with Child-Pugh A (score of 5 to 6)
  Interventions: Drug: JDQ443
- Moderate hepatic impairment (Experimental): Moderate hepatic impairment with Child Pugh B (score from 7 to 9)
  Interventions: Drug: JDQ443
- Severe hepatic impairment (Experimental): Severe hepatic impairment with Child Pugh C (score from 10 to 15)
  Interventions: Drug: JDQ443

INTERVENTIONS:
Drug: JDQ443 — All the participants will receive a single oral dose of JDQ443.

SUMMARY:
The purpose of this study is to evaluate the effect of hepatic impairment on the systemic pharmacokinetics (PK), safety, and tolerability of JDQ443 in participants with varying degrees of hepatic impairment.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, single-dose, multi-center, parallel group study to evaluate the PK of oral JDQ443 in participants with mild, moderate, and/or severe hepatic impairment compared to matched healthy control participants.

The study comprises a 28-day Screening period (Days -28 to -2), a baseline evaluation period (Day -1), a single dose administration of 200 mg of JDQ443 (Day 1), and a follow-up period of 4 days (Days 2 to 4) for PK sample collection. All participants should have a post-study safety follow-up contact conducted approximately 30 days after last administration of study treatment. The study will be considered complete once all the participants have finished the required assessments or have dropped out or been lost to follow-up.

A total of up to 48 participants will be enrolled in this study. Approximately 8 participants will be enrolled in each of mild (Child-Pugh A; Group 2), moderate (Child-Pugh B; Group 3), and severe (Child-Pugh C; Group 4) hepatic impairment groups (to have at least six evaluable participants in each group). Each participant in the healthy control group (Group 1) will be matched to one or more evaluable participants with hepatic impairment with respect to age, body weight and sex. All participants will receive a single JDQ443 dose. Upon completion of mild and moderate impairment groups, as well as matching control participants, an interim analysis will be conducted to compare the PK exposure of the two hepatic impaired groups (Groups 2 and 3) to that of the control participants. The interim analysis is to mitigate the potential safety risks in participants with severe hepatic impairment. If the interim analysis results do not show a clinically relevant increase in exposure of JDQ443 and is well tolerated from a safety perspective, then severe hepatic impairment participants may be enrolled. Participants with severe hepatic impairment will be enrolled only after the completion of the interim analysis.

ELIGIBILITY:
Key inclusion Criteria:

* Written informed consent must be obtained before any assessment is performed.
* Participants must weigh at least 50.0 kg to participate in the study and must have a body mass index (BMI) within the range of 18 to 40 kg/m2.
* Ability to communicate well with the investigator, to understand and comply with the requirements of the study.
* Participant must be willing to remain in the clinical research unit as required by the protocol.

Key exclusion Criteria:

* Use of other investigational drugs within the last 30 days or 5 half-lives prior to dosing, whichever is longer.
* Use of drugs (prescription, non-prescription and herbal remedies such as St John's wort) known to affect cytochrome p (CYP)3A, including both strong and moderate inhibitors and inducers, within 2 weeks prior to dosing until completion of the EOS Visit.
* Contradiction or hypersensitivity to the investigational compound/compound class or its excipients being used in this study.
* Pregnant or nursing (lactating) women. Pregnancy is defined as the state of a female after conception and until termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test.
* Known history of, or current clinically significant arrhythmias, history of prolonged QT correction formula (QTcF) interval or QTcF >480 msec

Other inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-05-03 (Actual); Primary Completion 2024-04-07 (Actual); Study Completion 2024-04-07 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-time Curve From Time Zero to the Last Quantifiable Concentration (AUClast) of JDQ443 | Day 1 (Pre-dose), 0.5, 1, 1.5, 2, 3 , 4 , 6 , 8 , 12 , 24 , 36 , 48 and 72 hours post-dose
  Blood samples will be collected for pharmacokinetics characterization. AUClast will be calculated from plasma concentration-time data using non-compartmental methods and summarized using descriptive statistics.
Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUCinf) of JDQ443 | Day 1 (Pre-dose), 0.5, 1, 1.5, 2, 3 , 4 , 6 , 8 , 12 , 24 , 36 , 48 and 72 hours post-dose
  Blood samples will be collected for pharmacokinetics characterization. AUCinf will be calculated from plasma concentration-time data using non-compartmental methods and summarized using descriptive statistics.
Maximum Observed Plasma Concentration (Cmax) of JDQ443 | Day 1 (Pre-dose), 0.5, 1, 1.5, 2, 3 , 4 , 6 , 8 , 12 , 24 , 36 , 48 and 72 hours post-dose
  Blood samples will be collected for pharmacokinetics characterization. Cmax will be calculated from plasma concentration-time data using non-compartmental methods and summarized using descriptive statistics.
Time to Reach the Maximum Concentration of JDQ443 After Drug Administration (Tmax) of JDQ443 | Day 1 (Pre-dose), 0.5, 1, 1.5, 2, 3 , 4 , 6 , 8 , 12 , 24 , 36 , 48 and 72 hours post-dose
  Blood samples will be collected for pharmacokinetics characterization. Tmax will be calculated from plasma concentration-time data using non-compartmental methods based on the actual time of sample collection and summarized using descriptive statistics
Time of observation prior to the first observation with a measurable concentration (Tlag) of JDQ443 | Day 1 (Pre-dose), 0.5, 1, 1.5, 2, 3 , 4 , 6 , 8 , 12 , 24 , 36 , 48 and 72 hours post-dose
  Blood samples will be collected for pharmacokinetics characterization. Tlag will be calculated from plasma concentration-time data using non-compartmental methods and summarized using descriptive statistics.
Terminal Elimination Half-life (T1/2) of JDQ443 | Day 1 (Pre-dose), 0.5, 1, 1.5, 2, 3 , 4 , 6 , 8 , 12 , 24 , 36 , 48 and 72 hours post-dose
  Blood samples will be collected for pharmacokinetics characterization. T1/2 will be calculated from plasma concentration-time data using non-compartmental methods and summarized using descriptive statistics.
Apparent Total Body Clearance From Plasma (CL/F) of JDQ443 following Drug Administration | Day 1 (Pre-dose), 0.5, 1, 1.5, 2, 3 , 4 , 6 , 8 , 12 , 24 , 36 , 48 and 72 hours post-dose
  Blood samples will be collected for pharmacokinetics characterization. CL/F will be calculated from plasma concentration-time data using non-compartmental methods and summarized using descriptive statistics.
Apparent Volume of Distribution of JDQ443 during Terminal Phase (Vz/F) | Day 1 (Pre-dose), 0.5, 1, 1.5, 2, 3 , 4 , 6 , 8 , 12 , 24 , 36 , 48 and 72 hours post-dose
  Blood samples will be collected for pharmacokinetics characterization. Vz/F will be calculated from plasma concentration-time data using non-compartmental methods and summarized using descriptive statistics.
Area Under the Plasma Concentration-time Curve from Time Zero to time "t" (AUC0-t) of JDQ443 | Day 1 (Pre-dose), 0.5, 1, 1.5, 2, 3 , 4 , 6 , 8 , 12 , 24 , 36 , 48 and 72 hours post-dose
  Blood samples will be collected for pharmacokinetics characterization. AUC0-t will be calculated from plasma concentration-time data using non-compartmental methods and summarized using descriptive statistics.
Latest pharmacokinetic sampling time with a measurable concentration (Tlast) of JDQ443 | Day 1 (Pre-dose), 0.5, 1, 1.5, 2, 3 , 4 , 6 , 8 , 12 , 24 , 36 , 48 and 72 hours post-dose
  Blood samples will be collected for pharmacokinetics characterization. Tlast will be calculated from plasma concentration-time data using non-compartmental methods and summarized using descriptive statistics.

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of unbound JDQ443 | Day 1 (Pre-dose), 0.5, 1, 1.5, 2, 3 , 4 , 6 , 8 , 12 , 24 , 36 , 48 and 72 hours post-dose
  Blood samples will be collected for pharmacokinetics characterization. Cmax of unbound drug will be calculated from plasma concentration-time data using non-compartmental methods and summarized using descriptive statistics.
Area Under the Plasma Concentration-time Curve From Time Zero to the Last Quantifiable Concentration (AUClast) of unbound JDQ443 | Day 1 (Pre-dose), 0.5, 1, 1.5, 2, 3 , 4 , 6 , 8 , 12 , 24 , 36 , 48 and 72 hours post-dose
  Blood samples will be collected for pharmacokinetics characterization. AUClast of unbound drug will be calculated from plasma concentration-time data using non-compartmental methods and summarized using descriptive statistics.
Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUCinf) of unbound JDQ443 | Day 1 (Pre-dose), 0.5, 1, 1.5, 2, 3 , 4 , 6 , 8 , 12 , 24 , 36 , 48 and 72 hours post-dose
  Blood samples will be collected for pharmacokinetics characterization. AUCinf of unbound drug will be calculated from plasma concentration-time data using non-compartmental methods and summarized using descriptive statistics.
Area Under the Plasma Concentration-time Curve From Time Zero to time "t" (AUC0-t) of unbound JDQ443 | Day 1 (Pre-dose), 0.5, 1, 1.5, 2, 3 , 4 , 6 , 8 , 12 , 24 , 36 , 48 and 72 hours post-dose
  Blood samples will be collected for pharmacokinetics characterization. AUC0-t of unbound drug will be calculated from plasma concentration-time data using non-compartmental methods and summarized using descriptive statistics.
Apparent Total Body Clearance From Plasma (CL/F) of unbound JDQ443 | Day 1 (Pre-dose), 0.5, 1, 1.5, 2, 3 , 4 , 6 , 8 , 12 , 24 , 36 , 48 and 72 hours post-dose
  Blood samples will be collected for pharmacokinetics characterization. CL/F of unbound drug will be calculated from plasma concentration-time data using non-compartmental methods and summarized using descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- United States (2):
  - Orlando Clinical Research Center, Orlando, Florida
  - Texas Liver Institute, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Link to study results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18281
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2550